CLINICAL TRIAL: NCT02621697
Title: Dual Task in Institutionalized Elderly: Positive Impact on the Risk of Falls and Functionality
Brief Title: Dual Task in Institutionalized Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Triangulo Mineiro (Other)
Responsible Party: Principal Investigator, Lislei Jorge Patrizzi, Phd, Universidade Federal do Triangulo Mineiro
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFTM 2015
Record Dates: First submitted 2015-08-14; First posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Aging
Keywords: dual task; aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive motor training (Experimental): Evaluate the effectiveness of a 12-week training based on dual-task (motor and cognitive) in institutionalized elderly.
  Interventions: Other: Cognitive motor training
- Control Group (Active Comparator): kinesiotherapeutic conventional treatment
  Interventions: Other: kinesiotherapeutic conventional treatment

INTERVENTIONS:
Other: Cognitive motor training — Initially an intervention consisting of double duty activities (motor-cognitive) and the control group will be subjected to a conventional treatment based on stretching and strengthening will be held.
  Arms: Cognitive motor training
Other: kinesiotherapeutic conventional treatment — Standardized global stretching and strengthening with squat exercise, plantar flexion in foot and elbow flexion supporting body weight in the hands arranged on the wall
  Arms: Control Group

SUMMARY:
Objectives: To evaluate the effects of eight weeks of cognitive motor training (dual task) in the risk of falls, balance, independence in basic activities of daily living (BADL) and handgrip in institutionalized elderly.

Methods: The sample was divided in two groups: double task group (DTG), consists of five elderly, undergoing a training consists of motor and cognitive activities and control group (CG) consists of four seniors who underwent conventional kinesiotherapeutic training, based on global stretching and strengthening exercises, both held in 16 sessions.

DETAILED DESCRIPTION:
Experimental, prospective and quantitative study, whose sample was selected for convenience in a long-term care institution for the elderly (LTCF) in the city of Uberaba - MG. The volunteers were divided into two groups, named dual task group (DTG) consists of five seniors, and control group (CG) consists of four elderly. All participants of both groups answered a questionnaire with sociodemographic and economic characteristics of the sample. Participants underwent a pre- and post evaluation containing vital signs parameters (blood pressure, respiratory rate and heart rate), anthropometric data (weight and height) and different tests to evaluate the balance, functional mobility, risk of falls, muscle strength and independence to carry out basic activities of daily living. The performed tests were Timed Up and Go (TUG) conventional, motor TUG and TUG cognitive, beyond Romberg test and Sensitized Romberg, Berg Balance Scale, and modified Katz scale (with maintenance of the six original activities of the scale, but with simulation to the performance of each task, measuring the spent time).

ELIGIBILITY:
Inclusion criteria:

* individuals over the age of 60,
* minimum score of 18 points on the Mini-Mental State Examination (MMSE),
* individuals classified as sedentary according the International Physical Activity Questionnaire (short version IPAQ-),
* literate and visual acuity preserved or corrected.

Exclusion criteria:

* Individuals unable to remain standing upright
* individuals dependent from auxiliary device to walk
* those who performed another type of physical therapy intervention concomitantly

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Risk of falls | 8 weeks of training
  Measured by the following tests: TUG, motor TUG, cognitive TUG, Romberg and sensitized Romberg (all measured in seconds)

SECONDARY OUTCOMES:
Independence to carry out basic activities of daily living | 8 weeks of training
  Through the modified Katz scale: the simulation of the activities originally present in the Katz scale was performed by the participants, and the time taken to their execution was recorded.
Muscle strength | 8 weeks of training
  Through dynamometry

CONTACTS AND LOCATIONS:
Overall Officials: Lislei Patrizzi, Professor, Principal Investigator — Universidade Federal do Triângulo Mineiro